CLINICAL TRIAL: NCT02199366
Title: Prospective Pilot Study of Early Markers of Radiation-Induced Cardiac Injury in Patients With Left-Sided Breast Cancer Receiving Photon or Proton Therapy
Brief Title: Study of Cardiac MRI in Patients With Left-Sided Breast Cancer Receiving Radiation Therapy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Ocala Royal Dames (Unknown)
Responsible Party: Sponsor
Other Study IDs: UFPTI 1419-BR02; IRB201800163 (Other: UF IRB); UFJ 2014-116 (Other: UF IRB Old Number)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Cardiac MRI; Radiation; Proton Radiation; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac magnetic resonance (cardiac MRI): Participants will have a cardiac MRI at baseline and within 1 year after completion of radiation therapy.
  Interventions: Procedure: Cardiac magnetic resonance (cardiac MRI)

INTERVENTIONS:
Procedure: Cardiac magnetic resonance (cardiac MRI) — Participants will have a cardiac MRI at baseline and within 1 year after completion of radiation therapy.
  Other Names: Cardiac MRI; CMR

SUMMARY:
This is a pilot study to determine if there are changes in heart function following completion of radiation therapy for breast cancer as measured by cardiac magnetic resonance imaging (cardiac MRI) scans. Additional purposes of this study are to assess cardiac side effects from radiation treatment, evaluate cardiac MRI changes by radiation technique, and compare quality of life questionnaires.

DETAILED DESCRIPTION:
As part of this study, participants will have a cardiac MRI at baseline and a follow-up cardiac MRI within 1 year after completion of standard radiation therapy for left-sided breast cancer. The cardiac MRI scans will be evaluated to determine if there are changes in cardiac function within 1 year after radiation treatment.

Patients will be asked to complete a questionnaire before and after treatment that asks about their health and any symptoms they may be having.

Physical exams and any other standard of care service or treatment will be at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Left-sided breast cancer stage I-III.
* Indications for adjuvant regional nodal and breast or chest wall radiation therapy (RT).
* Women and men are allowed.
* Must be at least 18 years old at time of consent.

Exclusion Criteria:

* Pregnant and/or breastfeeding women or patients of child-producing potential not willing to use contraception while on study.
* Prior history of cardiovascular disease per physician discretion.
* Stage 0 and IV breast cancer.
* Prior radiation therapy to chest.
* Concurrent trastuzumab per physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Radiation oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with changes in cardiac function. | 1 year after completion of radiation therapy
  A change in cardiac function may include shifts from baseline measures of LV mass, strain, ejection fraction, and late gadolinium enhancement.

SECONDARY OUTCOMES:
Proportion of patients with serious cardiac side effects. | 1 year after completion of radiation therapy
  Includes myocardial infarction, valve disorder, congestive heart failure, and angina.
Mean quality of life score. | 1 year after radiation treatment
  Comparison of baseline and post treatment quality of life questionnaires completed by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Bradley, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States